CLINICAL TRIAL: NCT02615353
Title: Preventing Diabetes in Latino Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Phoenix Children's Hospital (Other); St. Vincent de Paul Medical and Dental Clinic (Other); Valley of the Sun YMCA, Arizona (Other); University of Washington (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R01DK107579-01 (NIH); 3R01DK107579-03S1 (NIH)
Record Dates: First submitted 2015-11-04; First posted 2015-11-26 (Estimated); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Obesity; Diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle Intervention (Experimental): 6 months of a bi-weekly Nutrition Education, Physical Activity, and Behavioral Modification program
  Interventions: Behavioral: Intensive Lifestyle Intervention
- Usual Care Control (Placebo Comparator): Medical screening and dietary counseling with a Endocrinologist and Registered Dietitian
  Interventions: Other: Usual Care Control

INTERVENTIONS:
Behavioral: Intensive Lifestyle Intervention — 6-months of lifestyle education
  Arms: Lifestyle Intervention
Other: Usual Care Control — Medical visit and dietary counseling
  Other Names: Control
  Arms: Usual Care Control

SUMMARY:
Obesity and type 2 diabetes are critical public health issues in youth. This study will test the effects and estimate the cost-effectiveness of a culturally-grounded community-based lifestyle intervention on type 2 diabetes risk among obese Latino adolescents with prediabetes.

DETAILED DESCRIPTION:
Obesity and related health disparities represent some of the most significant public health challenges facing society. In particular, obese Latino adolescents are disproportionately impacted by insulin resistance and type 2 diabetes. Prediabetes is an intermediate stage in the pathogenesis of type 2 diabetes and represents a critical opportunity for intervention. The Diabetes Prevention Program established that lifestyle intervention can prevent or delay type 2 diabetes in adults with prediabetes. To date, no diabetes prevention studies have been conducted in obese Latino youth with prediabetes, a highly vulnerable and underserved group. Therefore, investigators propose a randomized-controlled trial to test the short-term (6-month) and long-term (12-month) efficacy of a culturally-grounded, lifestyle intervention, as compared to usual care, for improving glucose tolerance and reducing diabetes risk in 120 obese Latino adolescents with prediabetes. Investigators will further test intervention effects on changes in quality of life, explore the potential mediating effects of changes in total, regional, and organ fat on improving glucose tolerance and increasing insulin sensitivity, and estimate the initial incremental cost-effectiveness of the intervention as compared with usual care for improving glucose tolerance. The overall approach is framed within a multilevel Ecodevelopmental model that leverages community, family, peer, and individual factors during the critical transition period of adolescence when changes in health behaviors and health outcomes are linked to future health trajectories. The intervention is guided by Social Cognitive Theory and employs key behavioral modification strategies to enhance self-efficacy and foster social support for making and sustaining healthy behavior changes. The proposal builds upon extant collaborations of a transdisciplinary team of investigators working in concert with local community agencies to address critical gaps in how diabetes prevention interventions for obese Latino youth are developed, implemented and evaluated. This innovative approach is an essential step in the development of scalable, cost-effective, solution-oriented programs to prevent type 2 diabetes in this and other populations of high-risk youth.

ELIGIBILITY:
Inclusion Criteria:

* Latino: self-report
* Age: 12-16
* Obese: BMI percentile ≥95th percentile for age and gender or BMI ≥30 kg/m22
* Prediabetic: fasting glucose ≥100, or 2-hour post-OGTT glucose ≥120 mg/dl, or HbA1c ≥5.7

Exclusion Criteria:

* Taking medication(s) or diagnosed with a condition that influences carbohydrate metabolism, PA, and/or cognition
* Type 2 diabetes: Fasting glucose ≥126 mg/dl or 2-hour glucose ≥200 mg/dl, or HbA1c ≥6.5
* Recent Hospitalization (previous 2 months)
* Currently enrolled in (or within previous 6 months) a formal weight loss program.
* Diagnosed depression or other condition that may impact QoL

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 117 (Actual)
Dates: Start 2016-05-13 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Glucose Tolerance | 6-months, 12-months
  Change in 2 hour glucose concentration following a 75 gram Oral Glucose Tolerance Test
Insulin Sensitivity | 6-months, 12-months
  Change in Insulin Sensitivity following a 75 gram Oral Glucose Tolerance Test. Insulin sensitivity will be estimated by the Whole-body insulin sensitivity index (Matsuda Index).

SECONDARY OUTCOMES:
Youth Quality of Life | 6-months, 12-months
  YQOL has domains of self (feelings about one's self), social relationships (friends and family), environment (social and cultural milieu) are assessed and an overall QoL score is computed. The instrument shows strong psychometric properties including internal consistency (Chronbach's alpha >0.80), test-retest reliability (ICC >0.74), and construct validity with other pediatric QoL measures (r = 0.73, P<0.05 with KINDL). Weight specific QoL will be assessed by the YQOL-W which, measures three domains of weight-related QoL (Self, Social, and Environmental). It is specific to obese adolescents (11-18 years) for use in evaluating weight management interventions in clinical and community research. The instrument shows good reliability (ICC =0.77) and construct validity with the children's depression inventory (r=0.57, P<0.01) in adolescents and is more sensitive then generic measures for detecting changes in QoL among obese youth participating in lifestyle interventions.
Body Composition | 6-months, 12-months
  Change in fat mass and increase in lean tissue mass by DXA

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Soltero EG, Konopken YP, Olson ML, Keller CS, Castro FG, Williams AN, Patrick DL, Ayers S, Hu HH, Sandoval M, Pimentel J, Knowler WC, Frick KD, Shaibi GQ. Preventing diabetes in obese Latino youth with prediabetes: a study protocol for a randomized controlled trial. BMC Public Health. 2017 Mar 16;17(1):261. doi: 10.1186/s12889-017-4174-2. PMID 28302101
- [Derived] Pena A, Olson ML, Hooker E, Ayers SL, Castro FG, Patrick DL, Corral L, Lish E, Knowler WC, Shaibi GQ. Effects of a Diabetes Prevention Program on Type 2 Diabetes Risk Factors and Quality of Life Among Latino Youths With Prediabetes: A Randomized Clinical Trial. JAMA Netw Open. 2022 Sep 1;5(9):e2231196. doi: 10.1001/jamanetworkopen.2022.31196. PMID 36094502
- [Derived] Vander Wyst KB, Olson ML, Bailey SS, Valencia AM, Pena A, Miller J, Shub M, Seabrooke L, Pimentel J, Olsen K, Rosenberg RB, Shaibi GQ. Communicating incidental and reportable findings from research MRIs: considering factors beyond the findings in an underrepresented pediatric population. BMC Med Res Methodol. 2021 Dec 5;21(1):275. doi: 10.1186/s12874-021-01459-8. PMID 34865631
- [Derived] Vander Wyst KB, Olson ML, Hooker E, Soltero EG, Konopken YP, Keller CS, Castro FG, Williams AN, Fernandez ADR, Patrick DL, Ayers SL, Hu HH, Pena A, Pimentel J, Knowler WC, Shaibi GQ. Yields and costs of recruitment methods with participant phenotypic characteristics for a diabetes prevention research study in an underrepresented pediatric population. Trials. 2020 Aug 14;21(1):716. doi: 10.1186/s13063-020-04658-8. PMID 32799920